CLINICAL TRIAL: NCT01625247
Title: Drainage is Not Necessary Procedure After Laparoscopic Cholecystectomy Due to Severe Acute Cholecystitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2008-0140
Record Dates: First submitted 2012-06-12; First posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Acute Cholecystitis; Empyema
MeSH Terms: conditions — Cholecystitis, Acute; Empyema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 arm (Experimental): Patients under LC. Allocated to drain placement . Drainage was removed if the drainage amount was less than 20cc.
  Interventions: Procedure: Surgical drainage
- 2 arm (Active Comparator): Patients under LC. Allocation to sham drain,
  Interventions: Procedure: Surgical drainage

INTERVENTIONS:
Procedure: Surgical drainage — Postoperative abdominal drainage were connected to a 200-mL closed suction reservoir. The drainage was removed if there are drainage amount less than 20 mL and color was serous color.

SUMMARY:
Laparoscopic cholecystectomy (LC) is the current preferred method of cholecystectomy. The role of routine drainage after LC to decrease postoperative morbidity is still an issue of considerable debate. The goal of this study was to assess to role of drains in LC, performed for acute inflamed gallbladder.

ELIGIBILITY:
Inclusion Criteria:

* Acute cholecystis
* Laparoscopic cholecystectomy
* KAROFSKY PERFORMANCE SCALE > 70
* No history of major operation

Exclusion Criteria:

* NYHA class > 3
* Open cholecystectomy
* No- compliance
* Intraoperative injuries
* Inadequate hemostasis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
frequency of postoperative complication occurrence | whinin 1 week and 8 weeks postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance hospital, Seoul, Seoul, South Korea